CLINICAL TRIAL: NCT04914832
Title: Effectiveness of Covid-19 Vaccination in Eswatini Against SARS-CoV-2 Associated Hospitalization and Death
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shabir Madhi (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Shabir Madhi, Professor, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Eswatini Implementation & VE
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Pneumonia, Viral
Keywords: Vaccine; Effectiveness; COVID-19; pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Pneumonia | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Intervention Model Description: 1. Open-label, single-arm implementation study.
  2. Prospective hospital and mortuary-based case-control study with test-negative controls (test-negative case-control study) and other hospital controls (standard case-control study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All individuals who register on the National Vaccination Registry (Experimental): This will be open-label, single-arm implementation study in Eswatini. All individuals who register on the National Vaccination Registry will be eligible for enrolment. Participants will receive appointments for vaccination using the registry.
  Interventions: Biological: AZD1222

INTERVENTIONS:
Biological: AZD1222 — AZD1222 is a recombinant replication-defective chimpanzee adenovirus vaccine expressing the SARS-CoV-2 S surface glycoprotein.

SUMMARY:
Since late December 2019, the novel human coronavirus (SARS-CoV-2) first reported in China, has spread worldwide. Vaccines to prevent SARS-CoV-2 infections have been developed in record time and several candidate vaccines have completed Phase 2a/b and Phase 3 clinical trials.

Coronaviruses (CoVs) are spherical, enveloped viruses with positive-sense single-stranded RNA genomes. One fourth of their genome is responsible for coding structural proteins, such as the Spike (S) glycoprotein, envelope, membrane, and nucleocapsid proteins. Envelope, membrane, and nucleocapsid proteins are mainly responsible for virion assembly whilst the S protein is involved in receptor binding, mediating virus entry into host cells during CoVs infection via different receptors. SARS-CoV-2 belongs to the phylogenetic lineage B of the genus Betacoronavirus and it recognizes the ACE2 as the entry receptor. It is the seventh CoV known to cause human infections and the third known to cause severe disease after SARS-CoV and MERS-CoV.

AZD1222 is a recombinant replication-defective chimpanzee adenovirus vaccine expressing the SARS-CoV-2 S surface glycoprotein. Development of AZD1222, previously referred to as ChAdOx1 nCoV-19, was initiated by the University of Oxford, UK, with subsequent transfer of development activities to AstraZeneca. The ChAdOx1 platform has been used in 14 clinical studies sponsored by the University of Oxford with immunogens from multiple pathogens such as influenza, tuberculosis, malaria, chikungunya, Zika, MERS-CoV, and Meningitis B. Over 360 healthy adult participants have received ChAdOx1-vectored vaccines in these studies. These vaccines demonstrated robust immunogenicity after a single dose and favourable safety profiles, with no vaccine-related serious adverse events (SAEs).

DETAILED DESCRIPTION:
This will be open-label, single-arm implementation study in Eswatini. All individuals who register on the National Vaccination Registry will be eligible for enrolment. Participants will receive appointments for vaccination using the registry. Vaccination will be overseen by trained personnel. At enrolment participants will receive an intramuscular injection of AZ1222, a second dose will be given 10 weeks after the first injection. Surveillance for vaccine effectiveness will be performed at designated hospitals.

A prospective hospital-based, case-control study with test-negative controls (test-negative case-control design) and optionally other hospital controls (standard case-control design) will be conducted in parallel with the implementation study. Data will be collected through a network of hospitals located in Eswatini. A hospital-based case control study is an efficient design well suited to study for effectiveness against severe disease, and potentially allows for detailed medical information and additional data collection directly from the patient or healthcare provider. In addition, the study aims to determine the vaccine effectiveness (VE) of AZ1222 against severe disease due to the B.1.351 variant circulating in Southern Africa and other new variants that might evolve.

ELIGIBILITY:
Inclusion Criteria:

* Any individual aged 18 and older eligible to receive AZ1222 vaccine following the national immunization recommendations.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Any significant acute or chronic medical condition that in the opinion of the vaccinator makes the participant unsuitable for participation in the study or jeopardises the safety of the participant.
* Participant reports being pregnant.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the vaccine.

Test negative vaccine effectiveness case-control study

The study population consists of individuals presenting at the participating hospitals and health centres during the study period, who:

Either

* Are hospitalized (or died) for an illness consistent with possible COVID-19. Or (in case of other hospital controls)
* Presented to the emergency department (ED) for reasons other than a COVID-19 like illness (e.g. trauma or elective surgery).

And

* Meet the inclusion criteria.

Inclusion criteria:

* Ever eligible to receive AZ1222 vaccine following the national immunization recommendations prior to hospital admission.

And

* Willing and able to provide informed consent.

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75012 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of HIV-uninfected patients with laboratory-confirmed SARS-CoV-2 illness | 1 year
  Laboratory-confirmed SARS-CoV-2 illness (COVID-19) hospitalizations and deaths in HIV-uninfected individuals who have been vaccinated with at least 1 dose.
Number of patients with laboratory-confirmed SARS-CoV-2 illness who have been vaccinated with at least one dose | 1 year
  Laboratory-confirmed COVID-19 hospitalizations and deaths in individuals irrespective of HIV status [people living with (PLWH) and without HIV] who have been vaccinated with at least 1 dose.

SECONDARY OUTCOMES:
Number of HIV-uninfected patients with laboratory-confirmed SAR-CoV-2 illness | 1 year
  Laboratory-confirmed COVID-19 hospitalizations and deaths in HIV-uninfected individuals who have been fully vaccinated according to the national immunization recommendations.
Number of patients with laboratory-confirmed SARS-CoV-2 illness who have been fully vaccinated | 1 year
  Laboratory-confirmed COVID-19 hospitalizations and deaths in individuals irrespective of HIV status who have been fully vaccinated according to the national immunization recommendations.
Number of patients with laboratory-confirmed SARS-CoV-2 illness according to vaccination interval between doses | 1 year
  Laboratory-confirmed COVID-19 hospitalizations and deaths in individuals irrespective of HIV status who have been fully vaccinated according to the vaccine interval in between dose (≤4 weeks, 5-8 weeks, 8-11 weeks, ≥12 weeks).
Number of patients with laboratory-confirmed SARS-CoV-2 illness by genetic variant | 1 year
  The effect of AZD1222 vaccine on laboratory-confirmed COVID-19 hospitalizations and deaths in individuals irrespective of HIV status who have been vaccinated (with at least 1 dose/ fully vaccinated according to the national recommendations), by viral genetic variants (particularly B.1.351 and non-B.1.351 variants).
Number of patients of special interest with laboratory-confirmed SARS-CoV-2 illness | 1 year
  Laboratory-confirmed COVID-19 hospitalizations and deaths in individuals irrespective of HIV status who have been vaccinated (with at least 1 dose/ fully vaccinated according to the national recommendations), within populations of special interest (e.g. PLWH, specific age groups [special focus on the elderly], Chronic Respiratory Disease, Chronic Cardiovascular Disease, Chronic Kidney Disease, Chronic Liver Disease, Chronic neurologic Disease, Auto-Immune Disease, pregnant women, immunocompromised or specific chronic conditions).
Number of patients with laboratory-confirmed SARS-CoV-2 illness by time since vaccination | 1 year
  The effect of AZD1222 vaccine against laboratory-confirmed COVID-19 hospitalization and death in individuals irrespective of HIV status who have been vaccinated (with at least 1 dose/ fully vaccinated according to the national recommendations), by time since vaccination, including ≤14 days prior to symptom onset.

OTHER OUTCOMES:
Number of patients with laboratory-confirmed SARS-CoV-2 illness by level of disease severity | 1 year
  The AZD1222 vaccine effectiveness against laboratory-confirmed COVID-19 hospitalization and death in individuals irrespective of HIV status who have been vaccinated (with at least 1 dose/ fully vaccinated according to the national recommendations/ fully vaccinated according to the vaccine label), by level of severity. Three mutually exclusive categories: (i) hospital admission without intensive care unit (ICU) admission and without in-hospital death, (ii) ICU admission without in hospital death and (iii) in-hospital death.
Number of days in hospital among patients with laboratory-confirmed SARS-CoV-2 illness | 1 year
  To estimate the AZD1222 vaccine effect among laboratory-confirmed COVID-19 patients (vaccinated with at least 1 dose/ fully vaccinated according to the national recommendations) on the length of hospital stay (in days).
Number of patients with laboratory-confirmed SARS-CoV-2 illness stratified by SARS-CoV-2 seropositivity status | 1 year
  To estimate the AZD1222 vaccine effectiveness against laboratory-confirmed COVID-19 hospitalization and death in individuals irrespective of HIV status who have been vaccinated (with at least 1 dose/ fully vaccinated according to the national recommendations), stratified by SARS-CoV-2 seropositivity status (based on N-protein IgG) at admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Vaccination Center, Mbabane, Eswatini

REFERENCES:
- [Background] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298
- [Background] Greaney, A. J., A. N. Loes, K. H. D. Crawford, T. N. Starr, K. D. Malone, H. Y. Chu and J. D. Bloom (2021).
- [Background] Tegally H, Wilkinson E, Giovanetti M, Iranzadeh A, Fonseca V, Giandhari J, Doolabh D, Pillay S, San EJ, Msomi N, Mlisana K, von Gottberg A, Walaza S, Allam M, Ismail A, Mohale T, Glass AJ, Engelbrecht S, Van Zyl G, Preiser W, Petruccione F, Sigal A, Hardie D, Marais G, Hsiao NY, Korsman S, Davies MA, Tyers L, Mudau I, York D, Maslo C, Goedhals D, Abrahams S, Laguda-Akingba O, Alisoltani-Dehkordi A, Godzik A, Wibmer CK, Sewell BT, Lourenco J, Alcantara LCJ, Kosakovsky Pond SL, Weaver S, Martin D, Lessells RJ, Bhiman JN, Williamson C, de Oliveira T. Detection of a SARS-CoV-2 variant of concern in South Africa. Nature. 2021 Apr;592(7854):438-443. doi: 10.1038/s41586-021-03402-9. Epub 2021 Mar 9. PMID 33690265
- [Background] Volz, E., S. Mishra, M. Chand, J. C. Barrett, R. Johnson, L. Geidelberg, W. R. Hinsley, D. J. Laydon, G. Dabrera, Á. O'Toole, R. Amato, M. Ragonnet-Cronin, I. Harrison, B. Jackson, C. V. Ariani, O. Boyd, N. J. Loman, J. T. McCrone, S. Gonçalves, D. Jorgensen, R. Myers, V. Hill, D. K. Jackson, K. Gaythorpe, N. Groves, J. Sillitoe, D. P. Kwiatkowski, S. Flaxman, O. Ratmann, S. Bhatt, S. Hopkins, A. Gandy, A. Rambaut and N. M. Ferguson (2021).
- [Background] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Result] Fischer, R. J., N. van Doremalen, D. R. Adney, C. K. Yinda, J. R. Port, M. G. Holbrook, J. E. Schulz, B. N. Williamson, T. Thomas, K. Barbian, S. L. Anzick, S. Ricklefs, B. J. Smith, D. Long, C. Martens, G. Saturday, E. de Wit, S. C. Gilbert, T. Lambe and V. J. Munster (2021).